CLINICAL TRIAL: NCT06356506
Title: A Multicenter, Prospective Cohort Study on the Influencing Factors of Biochemical Response in Autoimmune Hepatitis
Brief Title: A Study on Factors of Biochemical Response in Autoimmune Hepatitis
Status: Not yet recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Xinyan, Director, Principal Investigator, Clinical Professor, Beijing Friendship Hospital
Other Study IDs: 2022-P2-338-01
Record Dates: First submitted 2024-01-22; First posted 2024-04-10 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Autoimmune Hepatitis
Keywords: Autoimmune hepatitis; Biochemical response; Prognosis; Immunosuppressive therapy
MeSH Terms: conditions — Hepatitis, Autoimmune

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, plasma, hemocyte, liver histopathology (if any)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Modeling group: The data of modeling group is used to construct a predictive model of AIH end-point events.
- Validation group: Validation group is used to validate the predictive model externally.

SUMMARY:
The goal of this observational study is to clarify the clinical characteristics of autoimmune hepatitis (AIH) in China. The main questions it aims to answer are:

Human leukocyte antigen (HLA) gene susceptibility in Chinese AIH patients prognostic factors associated with AIH Participants will provide liver tests results and details of treatment during follow-up.

DETAILED DESCRIPTION:
This study aims to establish a high-quality, standardized prospective cohort of AIH with regular follow-up, clarify the clinical characteristics of AIH in China, construct a prognostic model, and explore new serum markers or AIH gene susceptibility, so as to provide key clinical evidence for the prevention and treatment of AIH in China.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old at the time of onset;
2. AIH simplified score ≥6 and/or AIH revised score ≥10;
3. Liver biopsy was performed and consistent with the pathological diagnosis of AIH;
4. Patents were treatment naive or who were diagnosed and treated in other hospitals but have stopped glucocorticoid/immunosuppressive therapy for more than 3 months;
5. Agree to participate in this study and sign the informed consent form.

Exclusion Criteria:

1. concomitant liver diseases: hepatotropic viral hepatitis (A, B, C, D, and E) and non-hepatotropic viral hepatitis (cytomegalovirus and Epstein-Barr virus (EBV) infection);
2. concomitant with drug-induced liver injury, primary biliary cholangitis, primary sclerosing cholangitis, alcoholic liver disease, genetic and metabolic liver diseases;
3. bone marrow or liver transplantation;
4. incomplete baseline medical history and laboratory examination results;
5. for previously diagnosed patients, immunosuppressive therapy was discontinued less than 3 months;
6. Pregnancy or lactation;
7. patients with contraindications to glucocorticoid/immunosuppressive therapy;
8. complicated with other malignant tumors;
9. complicated with mental disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: AIH patients who fulfilled the inclusion and exclusion criteria were enrolled in this study.
Sampling Method: Probability Sample
Enrollment: 630 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2034-05-01 (Estimated); Study Completion 2034-05-01 (Estimated)

PRIMARY OUTCOMES:
Alanine aminotransferase (ALT) recovery | From time of enrollment to the date of first ALT recovery, assessed up to 120 months
  Normalization of ALT
Aspartate transaminase (AST) recovery | From time of enrollment to the date of first AST recovery, assessed up to 120 months
  Normalization of AST
Immunoglobulin G (IgG) recovery | From time of enrollment to the date of first IgG recovery, assessed up to 120 months
  Normalization of IgG
Death | From time of enrollment to the date of death from liver disease, assessed up to 120 months
  Patients die because of liver diseases
Liver transplantaiton | From time of enrollment to the date of liver transplantation, assessed up to 120 months
  Patients have liver transplantation because of AIH
Progression to hepatocellular carcinoma (HCC) | From time of enrollment to the first date of HCC diagnosed, assessed up to 120 months
  Patients progress to hepatocellular carcinoma due to poor treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Xinyan Zhao, Study Chair — Beijing Friendship Hospital; Zhengsheng Zou, Study Chair — Beijing 302 Hospital; Yu Chen, Principal Investigator — Beijing You 'an Hospital, Capital Medical University; Jia Li, Principal Investigator — Tianjin Second People's Hospital; Jingshou Chen, Principal Investigator — The First Affiliated Hospital of Xiamen University; Liang Wang, Principal Investigator — Lanzhou University Second Hospital; Huahua Wang, Principal Investigator — Jiaozuo People's Hospital; Xiaoli Hu, Principal Investigator — Heilongjiang Provincinal Hospital; Pingying Li, Principal Investigator — Qinghai People's Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No